CLINICAL TRIAL: NCT06286293
Title: YOD-RiSoCo: the Role of Social Cognition and Better Identification of Risk-taking Behaviour in Patients with Young-onset Dementia
Brief Title: YOD-RiSoCo: Social Cognition and Risk-taking Behaviour in Patients with Young-onset Dementia
Acronym: YOD-RiSoCo
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 18171
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-06

CONDITIONS: Young-onset Dementia
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- bvYOD: Neuropsychological assessment and driving simulator task.
  Interventions: Other: Neuropsychological assessment, driving simulator task
- non-bvYOD: Neuropsychological assessment and driving simulator task.
  Interventions: Other: Neuropsychological assessment, driving simulator task
- Patients with frontal brain damage: Neuropsychological assessment and driving simulator task.
  Interventions: Other: Neuropsychological assessment, driving simulator task
- Healthy controls: Neuropsychological assessment and driving simulator task.
  Interventions: Other: Neuropsychological assessment, driving simulator task

INTERVENTIONS:
Other: Neuropsychological assessment, driving simulator task — Neuropsychological assessment consisting of test measuring general cognitive abilities and social cognition. Driving simulator task measuring risk-taking.

SUMMARY:
The goal of this observational study is to learn about social cognition and risky behaviour in patients with young-onset dementia (YOD). The investigators want to

* Examine differences in performance on social cognition test and measures of risky behaviour between behavioural variant YOD patients, patients with frontal brain injury, non-behavioural YOD patients and healthy controls.
* Examine if there is a relation between social cognition tests and measures of risky behaviour.

Participants will be administered a neuropsychological assessment including social cognition measures and patients will complete a driving simulator task in which risky behaviour will be elicited.

ELIGIBILITY:
Inclusion Criteria:

All subjects

* Sufficient command of the Dutch language
* In possession of a driver's license with any driving experience throughout life
* Age 18 to 65

bvYOD subjects

* Probable diagnosis of young-onset dementia (before 65 years old), confirmed after interdisciplinary consensus meeting in which interviews, neuropsychological examination, neurological and psychiatric assessments, neuro-imaging, blood samples, and in some cases FDG/PIB-PETscans, CSF biomarkers or genetic counseling were discussed.
* Nosological diagnosis of bvFTD or bvAD

Non-bvYOD subjects

* Probable diagnosis of young-onset dementia (before 65 years old), confirmed after interdisciplinary consensus meeting in which interviews, neuropsychological examination, neurological and psychiatric assessments, neuro-imaging, blood samples, and in some cases FDG/PIB-PETscans, CSF biomarkers or genetic counseling were discussed.
* YOD subtypes other dan bvFTD or bvAD, such as amnestic variant AD.

Frontal brain injury subjects

- Neurological patients with frontal brain injury (e.g. traumatic brain injury, stroke or brain tumor patients).

Exclusion Criteria:

All subjects

* Suffering from severe motion sickness; motion sickness is a risk factor for simulator sickness

YOD subjects:

- Presence of premorbid severe neurological or psychiatric pathology, non-related to dementia.

Frontal brain injury subjects:

- Presence of serious psychiatric disorders or other neurological comorbidities.

Healthy control subjects:

* Presence of serious psychiatric disorders
* History of neurological disorders, which may interfere with cognitive functioning (e.g. recent concussion, previous subarachnoid or intracerebral haemorrhage, intracranial tumours, epilepsy, ischemic stroke).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with young-onset dementia, i.e. onset of dementia before the age of 65 years.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-02-04 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Social cognitive performance | 2024-2027
  Social cognition in bvYOD, compared to non-bvYOD, patients with frontal brain injury and healthy controls

SECONDARY OUTCOMES:
Association between social cognition and risky decision-making | 2024-2027
  Association between several aspect of social cognition (i.e. emotion recognition, empathy, theory of mind, emotion experience) and risk-taking behaviour.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gelmers F, Huitema RB, Scheenen ME, van Munster BC, Spikman JM; YOD-INCLUDED Consortium. Assessing social cognition and risk-taking behaviour in patients with young-onset dementia: Study protocol for the YOD-RiSoCo observational prospective cohort study. PLoS One. 2025 May 27;20(5):e0324517. doi: 10.1371/journal.pone.0324517. eCollection 2025. PMID 40424326